CLINICAL TRIAL: NCT01764685
Title: Topiramate to Reduce Heavy Drinking in HIV-Positive Heavy Drinkers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: We terminated the study due to problems recruiting alcoholic subjects with HIV.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Henry Kranzler, Professor of Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 816082
Record Dates: First submitted 2013-01-04; First posted 2013-01-09 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Heavy Drinking; HIV; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Topiramate; Practice Management, Medical

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topiramate + Medical Management (Experimental): Topiramate titrated up to 150 mg/day over 5 weeks then maintained for 6 weeks + Medical Management sessions for 15-25 minutes per study visit
  Interventions: Drug: Topiramate; Behavioral: Medical Management
- Placebo Pill + Medical Management (Placebo Comparator): Sugar pill with dosing schedule matched to intervention group + Medical Management sessions for 15-25 minutes per study visit
  Interventions: Behavioral: Medical Management; Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — Max therapeutic dose of 150mg/day
  Other Names: Topamax
  Arms: Topiramate + Medical Management
Behavioral: Medical Management — Medical Management (MM; Pettinati, 2004) will support patients' efforts to reduce their drinking. The study nurse makes direct recommendations for reducing drinking to sensible levels. The first session will use the brochure A Guide to Sensible Drinking (WHO 1996). The patient is provided with information about pharmacotherapy and the importance of adherence to topiramate/placebo. Subsequent treatment sessions (15-25 minutes) will be conducted at each study visit, during which the nurse will perform an assessment of the patient's drinking, monitor his/her medication adherence, and make recommendations to follow until the next visit. Men will be advised to consume no more than 2 drinks/day and 8 drinks/week; women will be advised to consume no more than 1 drink/day and 4 drinks/week.
Drug: Placebo — Placebo
  Arms: Placebo Pill + Medical Management

SUMMARY:
Heavy drinking (HD) is a risk factor for HIV transmission and is more common in HIV+ individuals than in the general population. HD adversely affects health directly and reduces adherence to antiretroviral therapies (ARTs), in part due to alcohol-induced cognitive impairment. Reduced drinking improves cognitive performance and adherence to ARTs. Medications approved in the United States to treat alcohol dependence have a small effect size. However, topiramate, FDA-approved as an anticonvulsant and a prophylaxis for migraine, has a greater effect size in reducing drinking and promoting abstinence in alcohol dependent individuals. To date, there are no studies of the effects of topiramate in HIV+ heavy drinkers. The investigators propose to conduct a randomized, parallel-groups, placebo-controlled, 11-week trial of topiramate in 40 HIV+ heavy drinkers who want to reduce or stop their drinking. There are three primary hypotheses for this feasibility and proof-of-concept study. First, the investigators hypothesize that topiramate-treated patients will decrease the frequency of their HD more than placebo-treated patients. Second, based on scores from computerized neurocognitive assessments, the investigators hypothesize that topiramate and placebo groups will show similar performance on a battery of cognitive tests. Third, based on self-reported medication adherence, the investigators hypothesize that adherence to ARTs will be greater in the topiramate group than in the placebo group. These findings will provide preliminary data to support a more definitive trial of topiramate for the treatment of HD in HIV+ heavy drinkers.

DETAILED DESCRIPTION:
A. General Design: This study will employ an 11-week, parallel-groups design (TOP vs. placebo) to test the effects of topiramate (TOP) on HD by HIV+ individuals with a current alcohol use disorder. We will gradually increase the dosage of TOP from 25 mg/day to 150 mg/day over a 6-week period to minimize adverse events. Random assignment to treatment group and double-blind conditions will be maintained throughout the study.

B. Recruiting: HIV+ men and women will be recruited through advertisements and by collaboration with physicians in the University of Pennsylvania Health System (UPHS) who will be invited to refer patients for whom heavy drinking in their HIV+ patients has created medical concerns. Patients will be recruited using the following methods: through referrals to the research center at the University of Pennsylvania (UPenn); by posting/distributing recruitment materials in community settings with public posting areas or other means of providing community access to materials (such as hospitals, town halls, public libraries, YMCA, health fairs/organizations); and through advertisements in local media (including text ads in newspapers, magazines; radio ads on local radio stations; web ads on internet sites and web postings on community message boards and research listings). These methods have been successful for Dr. Kranzler at the University of Pennsylvania and for many investigators at the Treatment Research Center (TRC) at UPenn. The TRC is an active center for clinical investigation and the staff and faculty there are highly experienced and capable in the conduct of clinical trials such as this. We will use institution-approved recruitment materials to advertise for regular or daily drinkers who are HIV+ and want to reduce their drinking. We will obtain permission at selected locations before distributing or posting the approved recruitment materials (to ensure that we comply with other institutions' guidelines). We anticipate that approximately 40% of patients will be women and that minority patients will be represented at least in proportion to the general population in Philadelphia. Based upon the large number of potential patients and our success in recruitment for prior studies, including those involving heavy drinkers, we are confident of our ability to achieve our recruitment goals.

C. Study Visits: At the screening visit, patients will provide informed consent and their reading ability will be evaluated, a medical and psychiatric history obtained. Blood and urine samples will be taken for routine clinical laboratory evaluations (including GGTP), drug screening, and pregnancy testing in females of reproductive potential. Patients will be interviewed with the Structured Clinical Interview for DSM-IV (SCID). Patients who are excluded will be referred to treatment.

The baseline visit will occur 1-14 days after the screening visit. Eligible patients will undergo a research evaluation, complete a packet of questionnaires, complete cognitive testing, and be interviewed by the research assistant. A physical examination will be performed by a study physician or nurse practitioner. Eligible patients will receive their first counseling session and first supply of study medication during a subsequent treatment session the same day. We will use urn randomization, a probabilistic balancing procedure to assign patients to medication group so that groups are balanced on key variables (Wei 1978): sex, race (white or non-white), number of HD days in past month.

During the 11-week treatment period, patients will return to the clinic weekly for five weeks while the dosage of the medication is gradually increased and then biweekly for six weeks. For patient safety during travel, they will be instructed not to drink prior to study visits. At each visit, the patient's breath alcohol level, weight, and vital signs will be measured. They will complete questionnaires and cognitive testing, and be interviewed by the research nurse about their use of concurrent medications, the occurrence of adverse events, and protocol compliance and then receive the medical management intervention. During visit 9 (end of treatment week 11), patients will complete questionnaires and cognitive testing and be interviewed by the research evaluator concerning their alcohol consumption. Patients will be compensated for this end-of-treatment visit. Patients will also be interviewed by the research nurse about their use of concomitant medications, occurrence of adverse events, compliance with the protocol, and their assessment of the effectiveness and acceptability of the treatment procedures (through the Medication Questionnaire; MED-Q). The nurse will dispense 4 days of medication for the taper and instruct the patient on how to take the medication during this period. Blood samples to measure serum GGTP will be obtained to assess the validity of self-reported drinking. A study nurse or research coordinator will call the patient one week after the endpoint visit to confirm that the subject completed the medication taper. Continuing adverse events will be followed by the study nurse and physician to their conclusion, as is feasible. Patients requesting (or clearly needing) additional treatment for alcohol problems will be referred to local treatment centers. All patients (including those who discontinue treatment prematurely) will be asked to complete an end-of-treatment evaluation and to complete all scheduled assessments to facilitate intention-to-treat (ITT) analyses. For patients who withdraw early and do not wish to continue with study visits/procedures, all end-of-treatment procedures will be administered at the time of withdrawal. Such patients will also be asked to undergo in-person or telephone follow-up at end-of-treatment for collection of the remaining treatment-phase Timeline Followback (TLFB) data.

D. Compensation: Patients will be compensated for their time and transportation.

E. Study Treatments: Throughout the study, we will maintain double-blind conditions with respect to medication administration. The research nurse, who is experienced in the conduct of alcohol pharmacotherapy trials, will deliver the medical management and monitor the medication, including capsule counts to measure adherence. The physician will meet with the patient initially, meet at least weekly with the nurse to discuss progress, and evaluate the patient in the event of severe or persistent adverse effects. The nurse will dispense study medications prescribed by the physician. Patients with severe psychological symptoms (e.g., suicidal thoughts) will be withdrawn from treatment and referred for appropriate clinical care. An effort will be made to obtain outcome information on all randomized patients for ITT analysis. In the medication condition, TOP will be administered at a maximum of 150 mg/day in two divided doses. TOP will be purchased commercially and formulated in opaque capsules by the Investigational Drug Service (IDS) at the University of Pennsylvania School of Medicine, which will purchase the TOP commercially and formulate the medication in capsules. Placebo will be formulated to match the active medication, such that inspection of the capsules will not permit the two to be differentiated.

F. Assessments:

Laboratory/Medical Assessments: These assessments are included to screen patients for medical exclusion criteria, assess potential adverse effects of medications, and corroborate self-reported drinking. Prior to entrance into the study, each patient will receive:

* A physical examination
* Urinalysis and urine toxicology
* Complete Blood Count (CBC)
* Gamma-Glutamyl Transferase Levels (GGTP)
* A chemistry panel (which includes electrolytes, liver enzymes, bilirubin, uric acid)
* Pregnancy testing in women of reproductive age (conducted at screening and then at the midpoint of the trial).

At the midpoint and end of the 11-week treatment phase, GGTP will be repeated to corroborate self-reported alcohol consumption. In addition to eliciting self-reported adverse events, weight and vital signs (blood pressure and pulse) will be obtained at each treatment visit.

Psychological/Behavioral Assessments:

* Sociodemographic information and alcohol dependence family history will be obtained at baseline.
* Locator information: At baseline, the research assistant will obtain information on patient locators nominated by the patient, which helps to maintain patients in treatment and enhances follow-up data collection.
* Psychiatric diagnosis: The Structured Clinical Interview(SCID-I/P; First et al. 2001) for the Diagnostic and Statistical Manual-IV (DSM-IV) will be used at baseline to classify patients according to the presence or absence of standard psychiatric disorders according to DSM-IV (American Psychiatric Association 1994).
* Alcohol use patterns and medication adherence: The Timeline Followback (TLFB; Sobell and Sobell 1992) will be used to estimate current medication adherence and alcohol consumption and drinking at intake and at each subsequent study visit. This interview procedure will provide quantity/frequency of alcohol consumption data for the period prior to the interview and since the last interview.
* Cogstate computerized battery: To examine the cognitive effects of changes in drinking behavior and of TOP treatment, we will administer the 20-minute battery biweekly. We will use these tasks: Detection Task, Identification Task, One Card Learning Task, One Back Memory Task, Shopping List Task, Groton Maze Learning Test.
* Iowa Gambling Task (IGT) (Decision Making and Impulsivity) [15 minutes]: The IGT (Bechara et al. 1994) is a computerized gambling task intended to simulate real-world decision making. Prior research indicates that it is sensitive to cognitive impairment in HIV populations (Martin et al. 2004) as well as substance users. Because practice effects are possible, the IGT will only be administered at baseline, midpoint (Visit 6), and endpoint (Visit 9).
* Depressive symptoms: Beck Depression Inventory (BDI)
* Medication adverse effects: Patients will provide subjective reports of adverse effects at each study visit using a list of adverse medication effects derived from completed studies of TOP for AD.
* Adherence to antiretroviral medication: We will use the Timeline Followback method to determine the percentage of ART doses taken each day as prescribed.
* Checklist of Cognitive Complaints: Individuals will rate their perceived impairment in everyday function in the domains of attention, memory, and decision making.
* General intellectual function: The Wechsler Test of Adult Reading (WTAR; Pearson Education, Inc.)
* Dementia screening: The Mini Mental State Exam (MMSE)

ELIGIBILITY:
Inclusion Criteria:

* Seropositive for HIV
* Age 18-70
* Report average of at least twice weekly heavy drinking
* Willing to reduce drinking to non-hazardous levels
* Verbal Intelligence Quotient (Verbal IQ) of 80 or higher
* Willing to provide signed informed consent
* Willing to nominate an individual to help locate the participant's whereabouts for follow-up
* If female: non-lactating and practicing a reliable method of birth control

Exclusion Criteria:

* Current clinically significant and/or uncontrolled physical disease (e.g., pancreatitis, diabetes)
* History of nephrolithiasis
* Severe psychiatric illness (i.e., psychosis or mania)
* Current diagnosis of drug abuse or dependence (other than nicotine abuse/dependence and cannabis abuse)
* Current diagnosis of alcohol dependence (AD) too severe for participation in a trial in which the goal is reduced drinking
* Gross cognitive impairment
* Glaucoma
* Serious/confounding neurological disease (e.g, stroke, seizure)
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry R. Kranzler, M.D., Principal Investigator — University of Pennsylvania; Kara R. Douglas, M.S., Study Director — University of Pennsylvania; Timothy S. Pond, M.P.H., Study Chair — University of Pennsylvania
Locations (1):
- University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Clinical research programs in the Department of Psychiatry at the Perelman School of Medicine/University of Pennsylvania — http://www.med.upenn.edu/psych/Programs.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate + Medical Management: Topiramate titrated up to 150 mg/day over 5 weeks then maintained for 6 weeks + Medical Management sessions for 15-25 minutes per study visit
  Topiramate: Max therapeutic dose of 150 mg/day
  Medical Management: (MM; Pettinati, 2004) will support patients' efforts to reduce their drinking. The study nurse makes direct recommendations for reducing drinking to sensible levels. The patient is provided with information about pharmacotherapy and the importance of adherence to topiramate/placebo. Subsequent treatment sessions (15-25 minutes) will be conducted at each study visit, during which the nurse will perform an assessment of the patient's drinking, monitor his/her medication adherence, and make recommendations to follow until the next visit. Men will be advised to consume no more than 2 drinks/day and 8 drinks/week; women will be advised to consume no more than 1 drink/day and 4 drinks/week.
Period: Overall Study
Arm/Group | Topiramate + Medical Management | Placebo Pill + Medical Management
Started | 0 | 4
Completed | 0 | 3
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Topiramate + Medical Management: Topiramate titrated up to 150 mg/day over 5 wks then maintained for 6 wks + Medical Management sessions for 15-25 mins per study visit
  Topiramate: Max therapeutic dose of 150mg/day
  Medical Management: Medical Management (MM; Pettinati, 2004) will support patients' efforts to reduce their drinking. The study nurse makes direct recommendations for reducing drinking to sensible levels. The first session will use the brochure A Guide to Sensible Drinking (WHO 1996). The patient is provided with information about pharmacotherapy and the importance of adherence to topiramate/placebo. Subsequent treatment sessions (15-25 mins) will be conducted at each study visit, during which the nurse will perform an assessment of the patient's drinking, monitor his/her medication adherence, and make recommendations to follow until the next visit. Men will be advised to consume no more than 2 drinks/day and 8 drinks/week; women will be advised to consume no more than 1 drink/day and 4 drinks/week.
- Total: Total of all reporting groups
Arm/Group | Topiramate + Medical Management | Placebo Pill + Medical Management | Total
Number analyzed (Participants) | 0 | 4 | 4
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 4 | 4
  >=65 years |  | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] |  | 50 [35 to 63] | 50 [35 to 63]
Gender [Number; unit: participants]
  Female |  | 0 | 0
  Male |  | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States |  | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Heavy Drinking Days Per Week by Medication Group
Description: Total number of heavy drinking days (>4 drinks for men; >3 drinks for women) for the placebo + medical management group during the study period. No data analysis will be done due to the small sample size and fact that all subjects received placebo study medication.
Time Frame: 11-week study period
Population: Data was only collected on 3 of the 4 subjects.
Measure: Number; unit: Number of heavy drinking days/week
Groups:
- Topiramate + Medical Management: Topiramate titrated up to 150 mg/day over 5 wks then maintained for 6 wks + Medical Management sessions for 15-25 mins per study visit
  Topiramate: Max therapeutic dose of 150mg/day
  Medical Management: Medical Management (MM; Pettinati, 2004) will support patients' efforts to reduce their drinking. The study nurse makes direct recommendations for reducing drinking to sensible levels. The first session will use the brochure A Guide to Sensible Drinking (WHO 1996). The patient is provided with information about pharmacotherapy and the importance of adherence to topiramate/placebo. Subsequent treatment sessions (15-25 minutes) will be conducted at each study visit, during which the nurse will perform an assessment of the patient's drinking, monitor his/her medication adherence, and make recommendations to follow until the next visit. Men will be advised to consume no more than 2 drinks/day and 8 drinks/week; women will be advised to consume no more than 1 drink/day and 4 drinks/wk.
Arm/Group | Topiramate + Medical Management | Placebo Pill + Medical Management
Number analyzed (Participants) | 0 | 3
Number of heavy drinking days/week |  | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 11 weeks each subject was enrolled in the study, the total study data was collected of 1 year.
Groups:
- Topiramate + Medical Management: Topiramate titrated up to 150 mg/day over 5 wks then maintained for 6 weeks + Medical Management sessions for 15-25 minutes per study visit
  Topiramate: Max therapeutic dose of 150mg/day
  Medical Management: Medical Management (MM; Pettinati, 2004) will support patients' efforts to reduce their drinking. The study nurse makes direct recommendations for reducing drinking to sensible levels. The first session will use the brochure A Guide to Sensible Drinking (WHO 1996). The patient is provided with information about pharmacotherapy and the importance of adherence to topiramate/placebo. Subsequent treatment sessions (15-25 minutes) will be conducted at each study visit, during which the nurse will perform an assessment of the patient's drinking, monitor his/her medication adherence, and make recommendations to follow until the next visit. Men will be advised to consume no more than 2 drinks/day and 8 drinks/week; women will be advised to consume no more than 1 drink/day and 4 drink
Arm/Group | Topiramate + Medical Management | Placebo Pill + Medical Management
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/4
Other Adverse Events (participants affected / at risk) | 0/0 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate + Medical Management (N=0) | Placebo Pill + Medical Management (N=4)
Increase in viral load from start to end of study (Immune system disorders) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Decrease in viral load from start to end of study (Immune system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
We closed our enrollment before meeting recruitment goals, due to difficulties with recruitment. We didn't analyze our data, due to a sample size of 4, that were all randomized to placebo group and only 3 of the 4 completed the study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No